CLINICAL TRIAL: NCT02107781
Title: A Prospective Observational Study of Continuous Intra-abdominal Pressure Monitoring in Patients With Postoperative Open Abdomen Undergoing Early Intervention and Closure
Brief Title: Intra-abdominal Pressure Monitoring in Patients With Open Abdomen Undergoing Early Closure
Status: Completed | Type: Observational
Sponsor: Michigan State University (Other)
Collaborators: ConvaTec Inc. (Industry)
Responsible Party: Principal Investigator, Benjamin Mosher, Assistant Professor, Department of Surgery, Michigan State University
Other Study IDs: r041998
Record Dates: First submitted 2014-01-24; First posted 2014-04-08 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Open Wound of Other and Unspecified Parts of Abdomen
Keywords: Open abdomen; abdominal compartment pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with open abdomen: Patients in a critical care unit with abdomen that was not closed during initial operation & will have intra-abdominal pressure monitoring using the AbViser abdominal compartment pressure measuring device.
  Interventions: Device: AbViser abdominal compartment pressure measuring device

INTERVENTIONS:
Device: AbViser abdominal compartment pressure measuring device — AbViser AutoValve IAP Monitoring Device will be used on all patient enrolled in the research study.
  Other Names: AbViser system; IAP system; Abdominal compartment syndrome monitor

SUMMARY:
The investigators will monitor the pressure generated inside the abdomen in a patient in whom the surgeon, for whatever reason, felt that the abdomen could not be closed at the initial operation. The investigators will aggressively treat rises in intra-abdominal pressure and see what changes, if any are found when the abdomen finally is closed.

DETAILED DESCRIPTION:
The detrimental effects of elevated intra-abdominal compartment pressure have been known for some time and are actively managed by most surgical critical care physicians. Similarly, it is well known that occasionally the abdomen cannot be immediately closed in some patients due to concern of elevated intra-abdominal pressure or ongoing contamination; these patients typically stay in hospital, often in expensive ICU's until final closure - and even then, some patients do not get definitive reconstruction of the abdominal wall until many months later, again adding to the expense of their care. Thus, there has been a move to give these patients early, aggressive closure of the abdomen, often using a combination of negative pressure wound therapy and biologic mesh. Currently these groups of patients who have early aggressive closure are incompletely studied; although abdominal compartment pressure measurements are routinely made on them, this is not commonly done intra-operatively when closure is being performed; nor have these patients been studied with continuous monitoring. This is especially striking considering the occlusive nature of negative wound therapy dressings: anecdotal increases in abdominal pressures have been noted in these patients, sometimes to dangerous levels. As there is accumulating evidence that diligent management of intra-abdominal pressure can improve outcomes in a variety of patients, there is an opportunity to apply accurate monitoring to a patient group that is also likely to benefit.

The investigators propose a prospective observational study on patients who are unable to be definitively closed at the time of surgery and are candidates for early aggressive abdominal closure. The investigators will monitor abdominal pressure using the AbViser continuous abdominal pressure monitoring device to ascertain whether there are episodes if intra-abdominal hypertension in these patients, and whether this improves or not after definitive closure. The research team will then attempt to correlate abdominal pressure measurements to outcomes. Finally the team will compare patients to historical controls using propensity scoring to explore differences in outcome.

Intra-abdominal pressure monitoring will be initiated when a patient has been identified as requiring an open abdomen. The monitoring will be done until the patient's abdominal wound has been closed and there are no elevated measurements. Once the patient has been discharged from the intensive care unit, the AbViser system will be discontinued. Patients will continue to be followed for the duration of their hospital stay and outcome measures will be assessed until discharge from the hospital, an expected average of 2 - 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Postoperative Surgical Patients who have not undergone abdominal closure, irrespective of the type of dressing used to protect the viscera

Exclusion Criteria:

* Age less than 18 years
* Coagulopathy
* Moribund/not expected to survive 48 hrs
* Patients in whom there is not a commitment to life supporting therapy
* Patients who have had definitive closure at the time of operation
* Patients in whom abdominal closure is not planned or not feasible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of patients in ICU with open abdomen
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2012-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Intra-abdominal pressure (IAP) Measurements | From the time when the patient has surgery & the abdomen is left open, immediately after abdomen is closed & until the patient's IAP system is discontinued, an expected average of 1 - 3 weeks.
  The IAP will be recorded using the AbVisor system when abdomen is open, after surgical closure and will continue until the IAP system is discontinued

SECONDARY OUTCOMES:
Length of time in critical care unit | From the time the patient is admitted to the critical care unit until discharged to a step-down unit. Measured immediately after discharge from critical care unit, an expected average of 1 - 3 weeks.
  The length of time subjects require monitoring in a critical care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D. Mosher, MD, Principal Investigator — Michigan State University
Locations (1):
- Sparrow Health System, Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: No